CLINICAL TRIAL: NCT00178334
Title: Screening for Urinary Incontinence by Primary Care Providers
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Gunhilde Buchsbaum, Associate Professor, University of Rochester
Other Study IDs: 11355
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to:

* Assess the rate of screening for urinary incontinence (UI) in women by their primary care providers
* Identify the type of screening used by primary care providers
* Identify barriers to screening for UI
* Identify differences in screening rates between specialties
* Assess whether primary care providers view UI as a serious medical problem
* Assess the comfort level of primary care providers in the diagnosis and treatment of UI
* Identify primary care providers' preferred mode of learning more about UI

DETAILED DESCRIPTION:
UI is a very common condition whose prevalence can be expected to increase dramatically in the coming decades. Treatment options are available to improve women's health and quality of life. However, inadequate communication between physicians and patients leads to decreased diagnosis and treatment. Past studies evaluating the use of screening by primary care providers, who act as gatekeepers in our healthcare system, clearly demonstrate that improvements must be made in the screening system. We propose a survey of local primary care providers to quantify screening rates for UI and identify barriers to successful screening. The information collected in this survey will allow us to identify methods such as targeted education opportunities and patient literature or questionnaires that will assist providers and their patients in initiating discussion and evaluation of UI.

ELIGIBILITY:
Inclusion Criteria:

* All primary care providers in the Greater Rochester metropolitan area, including: Primary care Medical Doctors (MD), Doctors of Osteopathy (DO), Primary care Nurse Practitioners (NP), and Physician Assistants (PA)

Exclusion Criteria:

* Physicians in the Greater Rochester metropolitan area who are not primary care providers

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care providers
Sampling Method: Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Response to mailing

CONTACTS AND LOCATIONS:
Overall Officials: Gunhilde Buchsbaum, MD, Principal Investigator — University of Rochester